CLINICAL TRIAL: NCT01257373
Title: Efficacy and Safety of Firebird 2 Cobalt-Chromium Alloyed Sirolimus-Eluting Stent in Treatment of Complex Coronary Lesions in Diabetes
Brief Title: Efficacy and Safety of Firebird 2 Stent in Treatment of Complex Coronary Lesions in Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Shanghai MicroPort Medical (Group) Co., Ltd. (Industry); CCheart Consulting Co., Ltd. (Industry)
Responsible Party: Wang Haichang, Department of Cardiology of Xijing Hospital , Fourth Military Medical University
Other Study IDs: XJ-2010-01
Record Dates: First submitted 2010-12-02; First posted 2010-12-09 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patiens with Firebird 2 stent: The group of 1300 patients, in which only Fireibrd2 stent is implanted, will be collected. All inclusive patients should be definitely diagnosed type 2 diabetic mellitus （DM）, either before or during the present hospitalization and with complex coronary lesion.
  Interventions: Device: Firebird 2 Cobalt-Chromium Alloyed Sirolimus-Eluting Stent

INTERVENTIONS:
Device: Firebird 2 Cobalt-Chromium Alloyed Sirolimus-Eluting Stent — Firebird2 CoCr-alloyed sirolimus-eluting stent system is the 2nd generation of drug-eluting stent(DES). It was registered successfully on Jan. 16, 2009 in China. This stent is based with a CoCr alloyed metal platform. The length is from 13-33mm, the diameter is from 2.5mm-4.0mm.

SUMMARY:
The goal of this study is to assess the long-term efficacy and safety of Firebird2 Cobalt-Chromium（CoCr）-alloyed sirolimus-eluting stent in treatment of complex lesions in diabetes.

DETAILED DESCRIPTION:
This clinical trial is an international multi-center prospective clinical registry research, for evaluating the efficacy and safety of Firebird 2 cobalt-chromium alloyed sirolimus-eluting stent in treatment of complex coronary lesions in diabetes. As planned, about 57 research centers all over China, Latin America and Asia-Pacific areas will be involved and, 1300 patients will be enrolled into this research. The implanted stents must all be Firebird2 cobalt-chromium alloyed sirolimus-eluting stent. The patient enrollment will last for 12 months. Clinical follow-up will be done respectively for 30 days, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months. All quitted patients during the study will not be replaced with any substitutes, but categorized in the enrollment failure column. The researcher must state clear the reason of nonenrollment.

ELIGIBILITY:
Inclusion Criteria:

* Definitely diagnosed type 2 DM either before or during the current hospitalization and with complex coronary lesions
* The coronary lesion is complied with the definition of complex type. (defined by protocol)
* The investigator admitted patients which are suitable for implanting Firebird2 CoCr-alloyed Sirolimus-eluting stent(SES)
* Patient or his/ her legal supervisor are provided with informed consents.

Exclusion Criteria:

* Women during pregnancy and breast-feeding;
* ST-segment elevated MI occurred within 1 week;
* Graft lesion after the coronary artery bypass graft(CABG) operation;
* Patient with other brand of stent implanted;
* LVEF ≤ 35%;
* Renal insufficiency before operation (Serum creatinine ≥ 177umol/L)
* Impaired fasting glucose（6.0mmol/L～7.0mmol/L）or impaired glucose tolerance（OGTT 2h blood glucose 7.8mmol/L～11.1mmol/L）patient;
* Recent PCI within 6 months or previous intravascular radiotherapy;
* Predicted life span is less than 12 months;
* Patient allergic to the following materials: aspirin, heparin, Clopidogrel, CoCr alloy, contrast agent or sirolimus.
* Recent participation of trial medication or other device study without endpoints completion or it is clinically interfering FIRE2-DIABETES study endpoints.
* Considered by other investigators unsuitable for implanting Firebird2 CoCr-alloyed SES
* Patients could not obey the study rules, such as not understanding the study manner, scope or its outcome, not cooperative, not providing the informed consent, not accepting follow-up, not finishing the whole study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry study will be conducted in 56 centers in which Firebird 2 stent is implemented. The data of 1300 patients, in which only Fireibrd2 stent is implanted, will be collected. All inclusive patients should be definitely diagnosed type 2 DM, either before or during the present hospitalization and with complex coronary lesions. The diagnosis criteria is the World Health Organization(WHO) recommended criteria 1999 version. I.e., fasting blood glucose ≥7.0mmol/L，random blood glucose ≥11.1mmol/L，or OGTT 2h blood glucose ≥11.1mmol/L. Impaired fasting glucose (6.0mmol/L～7.0mmol/L) or Impaired glucose tolerance (oral glucose tolerance test(OGTT) 2h blood glucose 7.8mmol/L～11.1mmol/L) can not be enrolled. The stress-induced hyperglycemia of acute coronary syndrome is illegible.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative major adverse cardiovascular events（MACE） | 12-month
  including cardiac death, Q-wave or Non-Q-wave MI,ischemia driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Post-procedure MACE | 30 days, 6/12/18/24/30/36 months.
Cumulative stent thrombosis | 12 months
  By Academic Research Consortium（ARC） definition (definite and probable)
Ischemia-driven target vessel revascularization(TVR) | 12 months
  The repeated intervention therapy or surgical bypass grafting to any segment of the target vessel is called target vessel revascularization. Target vessel means the entire major coronary arteries proximal or distal to the target lesion, including all upstream and downstream branches and the lesion itself
Stroke | 12 months
  including Ischemic and hemorrhagic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Haichang Wang, MD，PhD, Principal Investigator — Department of cardiology of Xijing Hospital, Fourth Military Medcical Univercsity
Locations (1):
- Department of cardiology of Xijing Hospital, Fourth Military Medical University, Xi'an, Shannxi, China